CLINICAL TRIAL: NCT01059890
Title: Cerebral Antibiotics Distribution After Acute Brain Injury
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Other Study IDs: A-BRAIN
Record Dates: First submitted 2010-01-29; First posted 2010-02-01 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Bacterial Infection; Brain Injury
MeSH Terms: conditions — Bacterial Infections; Brain Injuries | interventions — Cefotaxime; Metronidazole; Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cefotaxime (Experimental)
  Interventions: Drug: cefotaxime
- Metrodinazole (Experimental)
  Interventions: Drug: Metronidazole
- Ciprofloxacine (Experimental)
  Interventions: Drug: Ciprofloxacin
- Fosfocine (Experimental)
  Interventions: Drug: Fosfocine

INTERVENTIONS:
Drug: cefotaxime
  Arms: Cefotaxime
Drug: Metronidazole
  Arms: Metrodinazole
Drug: Ciprofloxacin
  Arms: Ciprofloxacine
Drug: Fosfocine
  Arms: Fosfocine

SUMMARY:
The aim of the study is to explore the distribution of antibiotics in the brain after an acute brain injury because brain infections treatment is still an health care problem.

ELIGIBILITY:
Inclusion Criteria:

* Acute brain injury
* Patient who receive an antibiotic for an infection or prophylaxy
* Glasgow coma score < 8

Exclusion Criteria:

* Age < 18 years old
* Pregnant woman
* HCV, HIV, HBV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-09; Primary Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Poitiers University Hospital - 2 rue de la Milétrie - Réanimation chirugicale, Poitiers, France